CLINICAL TRIAL: NCT06553664
Title: The Efficacy of Long-Course Treatment Using Disposable Gastrointestinal Vibrating Capsule (Vibrabot Capsule) for Chronic Constipation
Brief Title: The Efficacy of Long-Course Treatment Using Vibrating Capsules for Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, jiangxuan, Professor, Beijing Tsinghua Chang Gung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Long-Course Treatment
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Functional Constipation
Keywords: Chronic Functional Constipation; Vibrating Capsule; Long-Course Treatment
MeSH Terms: interventions — Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial group (Experimental): Subjects in the trial group took Vibrabot capsules at least 7 weeks, doses ranging from 2 to 5 capsules orally per week.
  Interventions: Drug: Treat with Vibrabot capsules for at least 7 weeks

INTERVENTIONS:
Drug: Treat with Vibrabot capsules for at least 7 weeks — Subjects in the trial group took Vibrabot capsules at least 7 weeks, doses ranging from 2 to 5 capsules orally per week.

SUMMARY:
This is a single-center trial. It enrolled nine 18- to 85-year-old patients with chronic constipation to evaluate the efficacy of long-course treatment by using vibrating capsule (VC).

DETAILED DESCRIPTION:
This study was a single-center prospective, single-arm exploratory clinical trial. If a subject signs an Ethics Committee (EC)-approved study informed consent (ICF) that meets the inclusion criteria and does not meet any of the exclusion criteria, the subject is considered eligible for admission to the study.

After completing a baseline questionnaire on bowel movements over the most recent 2 weeks, participants took VC at least 7 weeks, doses ranging from 2 to 5 capsules orally per week. After completion of treatment, subjects entered a follow-up period for at least 8 weeks. During the study period, the subjects are required to keep an e-diary recording daily bowel movements (BMs), medication intake, and discomforts, and complete the Patient Assessment of Constipation Symptoms (PAC-SYM) and the Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaires every two weeks.

Subjects are not expected to change their diet or lifestyle during the study. If the subject has not had a bowel movement for three or more consecutive days, the subject is allowed to use another method of defecation to assist with defecation. Subjects are required to avoid antibiotics, probiotics, prebiotics, and proton pump inhibitors throughout their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85-year-old men and women.
* Patients with symptoms of constipation in the six months prior to treatment, with less than three complete spontaneous bowel movements (CSBM) per week over the last three months, along with at least one of the following symptoms in at least 25% of bowel movements: Straining during defecation; Lumpy or hard stools (Bristol stool types 1-2) in at least 25% of bowel movements; A sensation of incomplete evacuation in at least 25% of bowel movements; A sensation of anorectal obstruction/blockage in at least 25% of bowel movements; Manual maneuvers to facilitate defecation (e.g., digital evacuation, pelvic floor support) in at least 25% of bowel movements. Loose stools are rarely present without the use of laxatives; insufficient criteria for irritable bowel syndrome Criteria fulfilled for the last three months with symptom onset at least six months prior to diagnosis.
* Patients with constipation not caused by organic disease based on medical history and previous medical records.
* Patients who agree to participate in the trial and voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients who are not eligible for surgery or those who refuse any abdominal surgery.
* Patients with known or suspected gastrointestinal obstruction, stenosis, diverticula, bleeding, deformities, or fistulas.
* Patients allergic to polymer materials.
* Patients with cardiac pacemakers or gastrointestinal pacemakers.
* Patients with abdominal aortic aneurysm, gastrointestinal vascular diseases, ulcers, or bleeding tendencies.
* Patients with swallowing disorders.
* Patients with severe depression or anxiety, or severe acute gastrointestinal diseases.
* Patients with history of gastrointestinal surgery or surgeries altering gastrointestinal structure (excluding appendectomy) or patients who underwent gastrointestinal endoscopic submucosal dissection (ESD) in the past three months.
* Patients with severe hemorrhoids (grade 3-4 as defined by the American Society of Colon and Rectal Surgeons guidelines).
* Patients planning to undergo magnetic resonance imaging (MRI) in the near future.
* Pregnant women or planning to become pregnant.
* Any other conditions deemed unsuitable for participation by the investigators.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
The proportions of responders during the treatment period. | at least 7 weeks
  Responders are the subjects with an average increase of ≥1 complete spontaneous bowel movements (CSBMs) per week during the treatment period compared to the baseline period.

SECONDARY OUTCOMES:
The proportion of patients with complete spontaneous defecation (CSBM) ≥three times per week during the treatment period. | at least 7 weeks
  Evaluating the proportion of patients with complete spontaneous defecation (CSBM) ≥three times per week during the treatment period.
Number of mean weekly complete spontaneous bowel movements (CSBM). | at least 7 weeks
  The average number of complete spontaneous bowel movements per week for each patient during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Jiang, Professor, Principal Investigator — Beijing Tsinghua Changung Hospital
Locations (1):
- XuanJiang, Beijing, Beijing Municipality, China